CLINICAL TRIAL: NCT06777498
Title: Optimizing Dietary Fiber Eating Patterns to Prevent Obesity and Resulting Metabolic Disorders
Brief Title: The Precision Nutrition New York Study
Acronym: PNNY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB0147806; 7005865 (Other Grant/Funding Number: USDA NIFA Hatch)
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Body Composition Changes; Body Weight Changes
Keywords: dietary fiber; gut microbiome; gut microbiota; short-chain fatty acids; SCFAs; whole grains; fruits; vegetables
MeSH Terms: conditions — Body Weight Changes | interventions — Vegetables; Fruit

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel arms in the intervention study. During each of the arms (pre and end time points), investigators will collect fecal samples and weigh the participants and measure body composition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group A: Whole grains then fruits and vegetables (Experimental): Whole grain intervention then fruits and vegetables
  Interventions: Other: Whole Grain Intervention then fruits and vegetables
- Experimental: Group B: Fruits and vegetables then whole grains (Experimental): Fruits and vegetables intervention then whole grains
  Interventions: Other: Fruit and Vegetable Intervention and then whole grains

INTERVENTIONS:
Other: Whole Grain Intervention then fruits and vegetables — TREATMENT 1: Participants will eat whole grains that add up to the required daily fiber needs. Investigators will provide participants with these products. Participants will follow this intervention for a set period of time. The beginning of the intervention will include a ramp up phase when they eat half of the daily fiber needs to prevent any gastrointestinal distress from suddenly consuming a higher fiber diet than usual.
  TREATMENT 2: Participants will eat fruits and vegetables that add up to the required daily fiber needs. Investigators will provide participants with these products. Participants will follow this intervention for a set period of time. The beginning of the intervention will include a ramp up phase when participants eat half of the daily fiber needs to prevent any gastrointestinal distress from suddenly consuming a higher fiber diet than usual.
  Arms: Experimental: Group A: Whole grains then fruits and vegetables
Other: Fruit and Vegetable Intervention and then whole grains — TREATMENT 1: Participants will eat fruits and vegetables that add up to the required daily fiber needs. Investigators will provide participants with these products. Participants will follow this intervention for a set period of time. The beginning of the intervention will include a ramp up phase when participants eat half of the daily fiber needs to prevent any gastrointestinal distress from suddenly consuming a higher fiber diet than usual.
  TREATMENT 2: Participants will eat whole grains that add up to the required daily fiber needs. Investigators will provide participants with these products. Participants will follow this intervention for a set period of time. The beginning of the intervention will include a ramp up phase when they eat half of the daily fiber needs to prevent any gastrointestinal distress from suddenly consuming a higher fiber diet than usual.
  Arms: Experimental: Group B: Fruits and vegetables then whole grains

SUMMARY:
Dietary fiber has been shown to have beneficial effects on human health through its impact on microbes present in the gut. However, these effects can vary between individuals, and everyone may not reap the same health benefits by eating the same sources of fiber. Factors predicting how an individual's gut microbes as well as the beneficial metabolites produced by these microbes change in response to different sources of fiber would be helpful in developing precision nutrition approaches that maximize the benefits of dietary fiber. The objective of this study is to evaluate candidate predictors of gut microbiota response to fiber sources from either whole grains or fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 21-50 years
* BMI is between 25-30. You can check your BMI here: https://www.cdc.gov/bmi/adult-calculator/index.html
* Must be able to have height, weight, waist, and hip circumference, and body composition measured during the study
* Must be able to provide saliva samples.
* Must be able to provide a phone number and email address at which the study investigators can contact for study-related matters.
* Must be able to increase dietary fiber intake to the recommended level following the instructions on the USDA MyPlate website: https://www.myplate.gov/myplate-plan
* Must be able to provide food records of everything consumed (food, beverage, and supplements) on one weekday and one weekend day (example Tuesday, Saturday) every week during the study. This will be done using an online survey.
* Must be able to provide 10 stool samples over 11 weeks of the study duration. 18) Must have stable weight (within ±3% of usual body weight) for the last two months.
* Must be able to to take an online survey to assess recent dietary fiber intake to determine eligibility.

Exclusion Criteria:

* Electronic medical implant, for example, a pacemaker.
* An existing, UNTREATED, thyroid condition.
* Use of systemic antibiotics (intravenous injection, intramuscular, or oral) within the last 4 months.
* An acute disease at the time of enrollment (Acute disease is defined as the presence of a moderate or severe illness with or without fever).
* A chronic, clinically significant (unresolved, requiring ongoing medical management or medication) pulmonary, cardiovascular, gastrointestinal, hepatic, or renal functional abnormality.
* Any suspected state of immunosuppression or immunodeficiency including HIV.
* A history of active UNTREATED gastrointestinal disorders or diseases including

  1. Inflammatory bowel disease (IBD)
  2. Ulcerative colitis (mild-moderate-severe)
  3. Crohn's or celiac disease
  4. Indeterminate colitis
  5. Irritable bowel syndrome (IBS) (moderate-severe)
  6. Persistent, infectious gastroenteritis, colitis or gastritis
  7. Persistent or chronic diarrhea of unknown etiology
  8. Clostridium difficile infection (recurrent)
  9. Chronic constipation
* Previously had bariatric surgery.
* An unstable dietary history as defined by major changes in diet during the previous month. For example, elimination or significantly increased intake of a major food group in the diet.
* Recent history of chronic alcohol consumption defined as more than 5 drinks (or servings) of alcohol per day.
* Female participants: pregnant/lactating.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight changes | 3-4 weeks
  For each intervention (whole grains & fruits and vegetables), investigators will measure change in body weight in kg = Post-intervention minus Pre-intervention
Body fat percentage changes | 3-4 weeks
  For each intervention (whole grains & fruits and vegetables), investigators will measure change in fat percentage = Post-intervention minus Pre-intervention

SECONDARY OUTCOMES:
Gut microbiome measured by 16S rRNA gene sequencing | 3-4 weeks
  For each intervention (whole grains & fruits and vegetables), investigators will calculate changes in relative abundance (proportion) of each gut bacterium from Pre-intervention to Post-intervention.
Fecal short-chain fatty acid concentrations (SCFAs) | 3-4 weeks
  For each intervention (whole grains & fruits and vegetables), investigators will measure change in SCFA concentrations = Post-intervention minus Pre-intervention. We will report the SCFAs acetate, butyrate, and propionate.

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell University, Ithaca, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will NEVER share de-identified data about the participants. Our previous publications show aggregated data results. This study is identical to our previous in design, sample types, and data being collected. We shared the de-identified 16S rRNA sequence data of the participants in a public database as requested by the journals. When requested by a journal, we have shared eligibility criteria. Some journals may require us to share our statistical code.